CLINICAL TRIAL: NCT00313443
Title: Study of Concentrations of Amiodarone in Fat Tissue Obtained by Needle Aspiration in Patients on Chronic Treatment
Brief Title: Concentrations of Amiodarone in Fat Tissue During Chronic Treatment
Acronym: ATACA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hopital Lariboisière (Other)
Collaborators: Unité de Recherches Therapeutiques - H. Lariboisiere (Unknown)
Responsible Party: Dr Carmelo Lafuente-Lafuente, Unité de Recherches Therapeutiques. Hopital Lariboisiere.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ATACA-URT04/06
Record Dates: First submitted 2006-04-10; First posted 2006-04-12 (Estimated); Results first posted 2009-08-06 (Estimated); Last update posted 2011-07-14 (Estimated); Status verified 2009-06

CONDITIONS: Arrhythmia; Atrial Fibrillation; Atrial Flutter
Keywords: Anti-Arrhythmia Agents; Amiodarone, chronic treatment; Amiodarone, adverse effects; Biopsy, Fine-Needle, Adipose tissue; Drug concentrations in tissues; Drug accumulation in tissues
MeSH Terms: conditions — Arrhythmias, Cardiac; Atrial Fibrillation; Atrial Flutter

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Amiodarone, long-term (Experimental): Unique arm: all patients were taking amiodarone for more than 6 months and all patietns underwent amiodarone dosage in blood and fat tissue samplings
  Interventions: Procedure: Fat tissue needle aspiration

INTERVENTIONS:
Procedure: Fat tissue needle aspiration — Small fat tissue sampling performed by needle aspiration.
  Other Names: Adipose subcutaneous tissue biopsy

SUMMARY:
The objective of this study is to determine if concentrations of amiodarone in fat tissue increases constantly over time during chronic treatment with this drug, and if blood concentrations reflect accurately the concentrations in fat tissue or not. This is because excessive concentrations of this drug in tissues can produce adverse effects.

DETAILED DESCRIPTION:
Amiodarone is very effective to treat cardiac arrhythmias but its use is limited by its toxicity, specially in chronic treatment. Accumulation of the drug in tissues is very probably the cause of the majority of amiodarone delayed adverse effects. However, this has not been proved because obtaining tissue samples is usually difficult and aggressive.

The investigators study, in patients following chronic treatment with amiodarone, if needle aspiration can provide samples of fat tissue useful to accurately determine amiodarone concentrations, how those concentrations in fat tissue correlate with cumulated dose, and how concentrations in fat tissue correlate with concentrations in blood, which is easier to obtain.

The investigators expect this knowledge will help to understand how amiodarone develops its adverse effects and possibly lead to new ways of monitoring treatment with this drug, or to adapt doses in chronic administration.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients taking amiodarone for more than 3 months (any dose, any indication)

Exclusion Criteria:

* Impossibility to perform needle aspiration of abdominal wall (local infection, skin disease)
* Coagulation disorders, INR > 3.0 if warfarin treatment
* Patient unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2006-04; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carmelo Lafuente-Lafuente, MD, Principal Investigator — Hopital Lariboisière, Internal Medicine "A" Service, Paris; Jean-Francois Bergmann, MD, Study Director — Hopital Lariboisiere, Internal Medicine "A" Service, Paris
Locations (1):
- Hopital Lariboisiere, Internal Medicine "A" and Cardiology Services, Paris, France

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment at a teaching hospital, from July 2006 to October 2007.
Pre-assignment Details: 67 consecutive patients were evaluated and 30 patients included. Reasons for non inclusion were: impossible to retrace history of amiodarone administration: 19 patients; less than 3 months on amiodarone treatment: 10 patients; unable to give informed consent: 4 patients; refused to participate: 4 patients.
Groups:
- Amiodarone/Fat Tissue Needle Aspiration: Unique arm: all patients underwent amiodarone dosage in blood and fat tissue samplings
Period: Overall Study
Arm/Group | Amiodarone/Fat Tissue Needle Aspiration
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Amiodarone/Fat Tissue Needle Aspiration
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 24
Age Continuous [Mean (Standard Deviation); unit: years] | 75 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 19
Region of Enrollment [Number; unit: participants]
  France | 30

OUTCOME MEASURES:

1. Primary Outcome: Relationship Between Amiodarone Concentration in Fat Tissue and Cumulated Dose.
Description: Correlation between amiodarone concentration in fat tissue (mean from several sampling points) and cumulated dose.
Time Frame: One single measure
Measure: Number; unit: Correlation coefficient R
Arm/Group | Amiodarone/Fat Tissue Needle Aspiration
Number analyzed (Participants) | 30
Correlation coefficient R | 0.20

2. Primary Outcome: Relationship Between Amiodarone Concentrations in Fat Tissue and in Plasma.
Description: Correlation between amiodarone concentrations in fat tissue (mean of 2 samples) and simultaneous concentration in plasma.
Time Frame: One single measure, taken just before daily administration
Measure: Number; unit: Correlation coefficient R
Arm/Group | Amiodarone/Fat Tissue Needle Aspiration
Number analyzed (Participants) | 30
Correlation coefficient R | 0.68

3. Primary Outcome: Relationship Between Amiodarone Concentrations in Fat Tissue and Developing Adverse Effects.
Description: Relationship between amiodarone concentrations in fat tissue (mean of two different samplings and developping adverse effects.
Time Frame: Cumulated time on amiodarone (varies in each patient)
Measure: Number; unit: Logistic regression OR
Arm/Group | Amiodarone/Fat Tissue Needle Aspiration
Number analyzed (Participants) | 30
Logistic regression OR | 1.01

4. Secondary Outcome: Pain and Complications (if Any) Caused by Fat Tissue Needle Aspirations
Description: Number of patients having complications (if any) caused by fat tissue needle aspirations
Time Frame: 24 hours after needle aspiration
Measure: Number; unit: Patients
Arm/Group | Amiodarone/Fat Tissue Needle Aspiration
Number analyzed (Participants) | 30
Patients | 2

5. Secondary Outcome: Presence of Any Adverse Effect Attributable to Amiodarone.
Description: Number of patients developing adverse effects by amiodarone leading to withdrawal or specific treatment (i.e. thyroid hormone treatment)
Time Frame: Cumulated time on amiodarone (varies in each patient)
Measure: Number; unit: Patients
Arm/Group | Amiodarone/Fat Tissue Needle Aspiration
Number analyzed (Participants) | 30
Patients | 11

ADVERSE EVENTS:
Arm/Group | Amiodarone/Fat Tissue Needle Aspiration
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 2/30
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Amiodarone/Fat Tissue Needle Aspiration (N=30)
Local Complications (if Any) Caused by Fat Tissue Needle Aspirations (Skin and subcutaneous tissue disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
Small number of patients included. High variability of amiodarone concentrations in fat tissue between the 2 simultaneous samples for some patients. Incidence of amiodarone-related adverse effects probably overestimated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No